CLINICAL TRIAL: NCT06904365
Title: Ovarian-Sparing Adaptive Radiotherapy in Young Adult Women (OvAR-Y): an In-Silico Feasibility Trial
Brief Title: Ovarian-Sparing Adaptive Radiotherapy in Young Adult Women
Acronym: OvAR-Y
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: 202502088
Record Dates: First submitted 2025-03-24; First posted 2025-04-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Uterine Cancer; Rectal Cancer; Colon Cancer; Breast Cancer; Lung Cancer; Sarcoma; Cervix Cancer; Head and Neck Cancer; Anal Cancer; Liver Cancer; Gastric Cancer; Bladder Cancer
Keywords: Young onset colorectal cancer; Early onset; Pre-menopausal; Ovarian sparing radiation
MeSH Terms: conditions — Uterine Neoplasms; Rectal Neoplasms; Colonic Neoplasms; Breast Neoplasms; Lung Neoplasms; Sarcoma; Uterine Cervical Neoplasms; Head and Neck Neoplasms; Anus Neoplasms; Liver Neoplasms; Stomach Neoplasms; Urinary Bladder Neoplasms | interventions — Radionuclide Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Ovarian-Sparing Adaptive Radiotherapy: A 25 Gy / 5 fx rectal plan for all patients, irrespective of their primary malignancy, will be created as per institutional standards. Patients may undergo treatment on any radiation therapy machine but will have their pelvis images on a HyperSight CBCT machine after consent while they receive their treatment. In general, patients will be imaged with 2 CBCTs approximately 10 minutes apart, each imaging session / day. However, only one CBCT per treatment session is required, and a patient may have between 1 to 10 scans total throughout 1 to 5 imaging sessions. In general, if ovaries are well visualized then only 1 or 2 imaging sessions will be completed.
  Interventions: Device: HyperSight cone beam computed tomography (CBCT) scan; Device: ETHOS 2.0

INTERVENTIONS:
Device: HyperSight cone beam computed tomography (CBCT) scan — HyperSight is a novel onboard imaging platform with a rapid-acquisition high-quality CBCT imager capable of acquiring images sufficient for simulation and treatment.
  Other Names: CBCT
Device: ETHOS 2.0 — ETHOS 2.0, an artificial intelligence treatment planning system, will be utilized in an emulator to create SCRT plans to determine the feasibility of clinically significant ovarian dose reductions in-silico.

SUMMARY:
Female patients with early onset (<50 years old) pelvic malignancies such as uterine and rectal cancers are rising in incidence, which often requires pelvic radiation; many of these patients are premenopausal and at a high risk of premature ovarian failure from radiotherapy. Premature ovarian failure carries significant cardiac, musculoskeletal, sexual, and psychosocial morbidity. Ovarian transposition carries variable success rates, is not readily accessible to the general population, and can still be at risk of clinically significant radiotherapy doses. There is an unmet need for innovative techniques to protect ovarian function.

ELIGIBILITY:
Inclusion Criteria:

* Biologic female
* Age between 18 and 50 years old (inclusive)
* Clinically premenopausal (defined as having active, regular menstruation without vasomotor symptoms)
* At least one of two ovaries readily visualized on diagnostic CT or MR imaging as confirmed by radiologist
* Planning to receive radiation therapy (for any indication)
* Ability to understand and willingness to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Prior pelvic radiation
* Prior cancer therapies that are known to impact ovarian function
* Prior diagnosis of ovarian insufficiency/failure or menopause
* Clinically peri- or post-menopausal

  * For patients > 45 years old, if there is a clinical history of vasomotor symptoms OR irregular periods, then the patient must be excluded.
  * For patients ≤ 45 years old, if there is a history of vasomotor symptoms consistent with menopause OR irregular menstruation for ≥3 months OR recent changes in their menstrual cycle > 14 days, then the patient must be excluded.
* Surgically removed or transposed ovaries
* Pregnant and/or breastfeeding

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will enroll patients at Siteman Cancer Center at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of ovarian visualization | Estimated to be 5 days
  Defined as being able to delineate at least one ovary (if only one is visible, must be the same ovary) for ≥60% of CBCT sessions per patient.

SECONDARY OUTCOMES:
Incidence of dosimetrically sparing one or both ovaries from a functionally ablative radiation dose | Estimated to be 5 days
  Defined as maintaining a cumulative >95% coverage of planned tumor volume (PTV) with 95% of the prescription dose (25 Gy/5 fx) while delivering no more 6 Gy to the ovaries per patient. If only one ovary can meet constraints it must be the same ovary over all fractions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Waters, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared if research proposal is submitted and approved by Principal Investigator.
Access Criteria: Email Principal Investigator with research proposal.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu